CLINICAL TRIAL: NCT00003854
Title: A Prognostic Study of Sentinel Node and Bone Marrow Micrometastases in Women With Clinical T1-2 N0 Breast Cancer
Brief Title: Prognostic Study of Sentinel Lymph Node and Bone Marrow Metastases in Women With Stage I or Stage IIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z0010; GUMC-00152; CDR0000067017 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunohistochemistry; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery + radiotherapy + adjuvant therapy (Experimental): Patients undergo bilateral anterior iliac crest bone marrow aspiration to test for presence of micrometastases. Patients then undergo breast-conserving therapy comprising segmental mastectomy and sentinel lymph node dissection (SLND) with planned postoperative whole-breast radiotherapy and systemic adjuvant therapy. The SLND comprises ipsilateral axillary sentinel node identification and histopathology.
  Patients with no sentinel node identified intraoperatively and patients with sentinel node metastasis identified by hematoxylin and eosin (H&E) who choose not to be registered to ACOSOG-Z0011 undergo axillary lymph node dissection involving removal of at least level I and II nodes.
  All patients undergo whole-breast radiotherapy (excluding a supraclavicular field) 5 days a week for a maximum of 8 weeks.
  Patients are followed at 30 days; at 6, 12, 18, 24, 30, and 36 months; and then annually until 10 years after surgery.
  Interventions: Other: immunohistochemistry staining method; Procedure: lymphangiography; Procedure: sentinel lymph node biopsy; Procedure: therapeutic conventional surgery; Radiation: whole breast irradiation

INTERVENTIONS:
Other: immunohistochemistry staining method
Procedure: lymphangiography
Procedure: sentinel lymph node biopsy
Procedure: therapeutic conventional surgery
Radiation: whole breast irradiation

SUMMARY:
RATIONALE: Biopsy of sentinel lymph nodes and bone marrow may improve the ability to detect and determine the extent of cancer.

PURPOSE: Phase III prognostic study of sentinel lymph node metastases and bone marrow metastases in women who have stage I or stage IIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the prevalence and evaluate the prognostic significance of sentinel lymph node micrometastases detected by immunohistochemistry in women with stage I or IIA breast cancer.
* Estimate the prevalence and evaluate the prognostic significance of bone marrow micrometastases detected by immunocytochemistry in these patients.
* Evaluate the hazard rate for regional recurrence in women whose sentinel nodes are negative by hematoxylin and eosin (H&E) staining.
* Provide a mechanism for identifying women whose sentinel nodes contain metastases detected by H&E so that these women can be considered as candidates for ACOSOG-Z0011.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be female.
2. Patient's clinical stage must be I or II (T1 or T2 N0 M0) and the tumor must be amenable to segmental mastectomy (lumpectomy).
3. Patient must have a tissue diagnosis of invasive breast carcinoma. Note: A patient can be registered to this study if they have a cytologic diagnosis suggestive of carcinoma from a fine needle aspiration (FNA) of a palpable or non-palpable breast lesion and the investigator believes the breast lesion is clinically suspicious for invasive breast carcinoma.
4. The date of the patient's first tissue diagnosis of invasive breast carcinoma or cytologic diagnosis of breast carcinoma must be no more than 60 days prior to SLND.
5. The patient who had segmental mastectomy (lumpectomy) performed previously, and is now referred to the local investigator for SLND, is eligible if the lumpectomy was less than or equal to 60 days prior to the SLND. Copies of the operative and pathology reports must be submitted as a part of the registration process.
6. Patient must have ECOG/Zubrod status of ≤2, as documented in patient's medical record.
7. Patient must be available for follow-up.
8. The patient with a history of a previous malignancy is eligible for this study as long as the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided that the following criteria are met:

   1. The patient has undergone potentially curative therapy for all prior malignancies.
   2. There has been no evidence of any prior malignancies for at least five years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone), and
   3. The patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.
9. Signed and dated informed consent is obtained prior to patient registration.
10. Patients of childbearing potential must have a negative serum or urine pregnancy test within 14 days of beginning study interventions.
11. Patient must be able to physically undergo bilateral anterior iliac crest bone marrow aspiration.

Exclusion Criteria:

1. Patient is lactating (breastfeeding).
2. Patient has been previously treated with chemotherapy, estrogen receptor antagonists (i.e. Tamoxifen) or selective estrogen receptor modulators (SERMs, i.e. Raloxifene) for this invasive breast cancer.
3. Patient has a previously placed pre-pectoral breast implant. NOTE: A subpectoral implant is allowed.
4. Patient is considered a poor surgical risk due to a non-malignant systemic disease (cardiovascular, renal, etc.), which would preclude the treatment options.
5. Patient has concurrent bilateral invasive breast malignancies.
6. Patient is not able to undergo and does not have access to radiation therapy as describedin Adjuvant Radiation Therapy in the Interventions section of the protocol.

   Patients with active connective tissue disorders and those that live too far from a radiation treatment center, for example, would not be eligible.
7. Patient has clinically and radiologically identified multi-centric disease that is not amenable to a single lumpectomy.
8. Patient has had previous ipsilateral axillary surgery such as excisional biopsy of lymph node(s), treatment of hidradenitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4590 (Actual)
Dates: Start 1999-04; Primary Completion 2006-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 10 years

SECONDARY OUTCOMES:
Disease-free survival | Up to 10 years
Axillary recurrence following detection of negative SN with H&E staining in women who did not have an ALND | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Armando E. Giuliano, MD, Study Chair — Saint John's Cancer Institute
Locations (116):
- United States (113):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital - Mobile AL, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - St. Vincent Doctors Doctors Hospital, Little Rock, Arkansas
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Summit Medical Center, Oakland, California
  - St. Joseph Hospital - Orange, Orange, California
  - Huntington Memorial Hospital, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - Donald N. Sharp Memorial Community Hospital, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Watson Clinic, Lakeland, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Martin Memorial Cancer Medical Center, Stuart, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - DeKalb Medical Center, Inc., Decatur, Georgia
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kaiser Permanente Medical Center, Honolulu, Hawaii
  - St. Luke's Regional Medical Center, Boise, Idaho
  - St. Elizabeth's Hospital, Belleville, Illinois
  - Belleville Memorial Hospital, Belleville, Illinois
  - Northwestern University Medical Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Little Company of Mary Hospital - Evergreen Park, Evergreen Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Anthony Memorial Health Center - Michigan City Campus, Michigan City, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Spectrum Health - Butterworth Campus, Grand Rapids, Michigan
  - Henry Ford Medical Center - West Bloomfield, West Bloomfield, Michigan
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Columbia Regional Hospital, Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Lester E. Cox Medical Centers, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Lutheran Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Kingston Hospital, Kingston, New York
  - Benedictine Hospital, Kingston, New York
  - St. Luke's-Roosevelt Hospital Center - Roosevelt Division, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Durham Regional Hospital, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Texas Cancer Center at Brackenridge Hospital, Austin, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - St. Paul University Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Carilion New River Valley Medical Center, Christiansburg, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Health System - Cancer Center of Western Virginia, Roanoke, Virginia
  - Columbia Lewis-Gale Medical Center, Salem, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Peter MacCallum Cancer Institute, East Melbourne, Victoria, Australia
- Ireland (2):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin

REFERENCES:
- [Background] Olson JA Jr, McCall LM, Beitsch P, Whitworth PW, Reintgen DS, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Giuliano AE; American College of Surgeons Oncology Group Trials Z0010 and Z0011. Impact of immediate versus delayed axillary node dissection on surgical outcomes in breast cancer patients with positive sentinel nodes: results from American College of Surgeons Oncology Group Trials Z0010 and Z0011. J Clin Oncol. 2008 Jul 20;26(21):3530-5. doi: 10.1200/JCO.2007.15.5630. PMID 18640934
- [Result] Hunt KK, Ballman KV, McCall LM, Boughey JC, Mittendorf EA, Cox CE, Whitworth PW, Beitsch PD, Leitch AM, Buchholz TA, Morrow MA, Giuliano AE. Factors associated with local-regional recurrence after a negative sentinel node dissection: results of the ACOSOG Z0010 trial. Ann Surg. 2012 Sep;256(3):428-36. doi: 10.1097/SLA.0b013e3182654494. PMID 22868365
- [Result] Giuliano AE, Hawes D, Ballman KV, Whitworth PW, Blumencranz PW, Reintgen DS, Morrow M, Leitch AM, Hunt KK, McCall LM, Abati A, Cote R. Association of occult metastases in sentinel lymph nodes and bone marrow with survival among women with early-stage invasive breast cancer. JAMA. 2011 Jul 27;306(4):385-93. doi: 10.1001/jama.2011.1034. PMID 21791687
- [Result] Wilke LG, Ballman KV, McCall LM, Giuliano AE, Whitworth PW, Blumencranz PW, Reintgen DS, Burak WE, Leitch AM, Hunt KK. Adherence to the National Quality Forum (NQF) breast cancer measures within cancer clinical trials: a review from ACOSOG Z0010. Ann Surg Oncol. 2010 Aug;17(8):1989-94. doi: 10.1245/s10434-010-0980-9. Epub 2010 Mar 23. PMID 20309640
- [Result] Wilke LG, McCall LM, Posther KE, Whitworth PW, Reintgen DS, Leitch AM, Gabram SG, Lucci A, Cox CE, Hunt KK, Herndon JE 2nd, Giuliano AE. Surgical complications associated with sentinel lymph node biopsy: results from a prospective international cooperative group trial. Ann Surg Oncol. 2006 Apr;13(4):491-500. doi: 10.1245/ASO.2006.05.013. Epub 2006 Mar 2. PMID 16514477
- [Result] Leitch AM, Beitsch PD, McCall LM, Posther K, Newman LA, Herndon JE 2nd, Hunt KK, Giuliano AE. Patterns of participation and successful patient recruitment to American College of Surgeons Oncology Group Z0010, a phase II trial for patients with early-stage breast cancer. Am J Surg. 2005 Oct;190(4):539-42. doi: 10.1016/j.amjsurg.2005.06.024. PMID 16164916
- [Result] Posther KE, McCall LM, Blumencranz PW, Burak WE Jr, Beitsch PD, Hansen NM, Morrow M, Wilke LG, Herndon JE 2nd, Hunt KK, Giuliano AE. Sentinel node skills verification and surgeon performance: data from a multicenter clinical trial for early-stage breast cancer. Ann Surg. 2005 Oct;242(4):593-9; discussion 599-602. doi: 10.1097/01.sla.0000184210.68646.77. PMID 16192820
- [Derived] Katz MS, McCall L, Ballman K, Jagsi R, Haffty BG, Giuliano AE. Nomogram-based estimate of axillary nodal involvement in ACOSOG Z0011 (Alliance): validation and association with radiation protocol variations. Breast Cancer Res Treat. 2020 Apr;180(2):429-436. doi: 10.1007/s10549-020-05555-z. Epub 2020 Feb 10. PMID 32043193